CLINICAL TRIAL: NCT04758572
Title: Effects of a Manual Therapy Program in Patients With Plantar Fasciitis
Brief Title: Efficacy of Manual Therapy in Plantar Fasciitis
Acronym: MTPlantarF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID0033
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Plantar Fasciitis
Keywords: pain; function; treatment
MeSH Terms: conditions — Fasciitis, Plantar; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy (Experimental): Mobilization. Axial decoaptation, talar mobilization, global and specific articulatory mobilization of the foot, mobilization of the fibular head, femorotibial mobilization, hip mobilization. In addition, lumbar joint mobilization is applied. It lasted 20 minutes. Subsequently, Trigger Point Inhibition is applied. in the medial gastrocnemius, soleus, and square plantar muscles.
  Plantar fascia massage. A deep friction technique was applied longitudinally and transversely to the plantar fascia and the triceps surae. The duration was 5/10 minutes Passive stretching. Stretches were applied to the plantar fascia, the gastrocnemius muscles and the soleus muscles in order to relax these muscles. The duration was 5/10 minutes.
  Interventions: Other: Manual Therapy
- Massage (Active Comparator): Consist of gentle kneading and rubbing based on a muscle chain protocol (20 minutes), and the same trigger point Inhibition, plantar fascia massage, and passive stretching.
  Interventions: Other: Massage muscle chain

INTERVENTIONS:
Other: Manual Therapy — Mobilization, massage and stretching
  Arms: Manual Therapy
Other: Massage muscle chain — Massage very soft following the directions of the muscle chains, massage and stretching
  Arms: Massage

SUMMARY:
Plantar fasciitis is characterized by localized pain at the insertion site of the plantar fascia on the calcaneus. The pain worsens in the morning with the first step of the foot, after resting or at the beginning of a workout, it can increase after intense activity and persist even when it stops. The first-line plantar fasciitis treatment is conservative. Although few studies have currently evaluated the effectiveness of physical therapy, it appears that the combination of several techniques is more effective than any technique used in isolation. The objective of this study is to know the results of two manual therapy treatments in terms of pain and functionality with a direct action on the plantar fascia.

Patients diagnosed with plantar fasciitis will be recruited. They will be randomly assigned into two intervention groups: Group 1 will receive a direct treatment on the plantar fascia and posterior aspect of the leg to relax and elongate the tissues. It will consist of manual therapy of the foot and ankle, treatment of the trigger points of the soleus muscle and plantar square, and also massage, and passive stretching and group 2 will receive a treatment with superficial massage based on a muscle chain protocol. It lasts 4 weeks, evaluations will be carried out at the beginning of treatment, at the end of the treatment and a follow-up one month. The evaluations will consist of pain on pressure, ankle goniometry, pain, lower limb functionality dynamic balance, function and daily activities and ankle ability scale.

DETAILED DESCRIPTION:
Introduction Plantar fasciitis is characterized by localized pain at the insertion site of the plantar fascia on the calcaneus, which can radiate toward the medial edge of the foot. The pain worsens in the morning with the first step of the foot, after resting or at the beginning of a workout, it can increase after intense activity and persist even when it stops. These symptoms can lead to functional limitation and prolonged disability. It is one of the most common foot pathologies. The first-line plantar fasciitis treatment is conservative. Although few studies have currently evaluated the effectiveness of physical therapy, it appears that the combination of several techniques is more effective than any technique used in isolation.

The objective of this study is to know the results of two manual therapy treatments in terms of pain and functionality with a direct action on the plantar fascia.

Material and methods

Patients diagnosed with plantar fasciitis will be recruited. Patients will sign an explanatory informed consent for the project before starting it. All patients are volunteers. They will be randomly assigned into two intervention groups:

* Group 1 will receive a direct treatment on the plantar fascia and posterior aspect of the leg to relax and elongate the tissues. It will consist of manual therapy of the foot and ankle, treatment of the trigger points of the soleus muscle and plantar square, and also massage, and passive stretching.
* Group 2 will receive a treatment with superficial massage based on a muscle chain protocol.

The intervention consists of a 4-week application, evaluations will be carried out at the beginning of treatment, at the end of the treatment and a follow-up one month.

The evaluations will consist of pain on pressure using an algometer, ankle goniometry, pain and lower limb functionality with the validated Foot Function Index scale, dynamic balance using the Star Excursion Balance Test, evaluation of the function and daily activities with the Foot and ankle ability scale.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old, diagnosed with plantar fasciitis.
* Evolution of fasciitis greater than 1 month
* Not being receiving any other type of physiotherapy treatment at the time of the study.

Exclusion Criteria:

* Subjects showing tumor, lower limb fractures, rheumatoid arthritis, vascular disease, administration of corticosteroids for long periods of time, pregnancy, previous surgeries in the affected or scheduled surgeries during the study period.
* Subjects who were not able to understand or respond to the evaluations of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Foot pain | 8 week
  Pressure pain threshold is measured by digital algometer to determine overall pressure pain sensitivity at which a sensation of pressure changed to pain. The patient is placed in a prone position with the feet off the table, gradual pressure is applied to the insertion area of the plantar fascia on the calcaneus with the algometer until the sensation of pressure becomes painful. The pressure (cm2/kg) is applied perpendicular to the skin at a speed of 30 kPa/s. Three measurements are applied, with 1 minute between them, and the average is recorded.

SECONDARY OUTCOMES:
Ankle flexion | 8 week
  Evaluation of passive ankle flexion is carried out using a universal goniometer. With the subject in the supine position and with the knees extended, the fulcrum of the goniometer is placed on the lateral malleolus, the mobile arm on the fifth metatarsal, and the fixed arm on the fibula.
Dynamic balance | 8 week
  Evaluation using the Star Excursion Balance Test (SEBT). Its purpose is the prediction of the risk of injury to the lower extremities and the identification of dynamic balance deficits. It is carried out in a standing position and with previous training, the subjects perform the test 4 times before their final evaluation. The subject must remain stable while performing movements of the lower limb in different directions (anterior, lateromedial, lateroposterior) while the other remains fixed and stable at one point.
Quality of life in relation to foot pain | 8 week
  It is evaluated using the SF-12 questionnaire. It is a questionnaire that assesses the quality of life of patients and is composed of 12 questions about the health of the participants and informs us about the physical (PCS) and mental (MCS) health of the subjects. The score ranges from 0 to 100.
Foot health | 8 week
  We will evaluate using the Foot Health Status Questionnaire (FHSQ) (25). It consists of three sections with a total of 23 items in total. Section 1 assesses foot function, foot pain, footwear, and general foot health, making up 13 of the 23 items. Section 2 assesses general health, physical activity, and social ability. Section 3 assesses the socioeconomic level, comorbidity and satisfaction.
Impact and disability from foot pain | 8 week
  Evaluation using the Foot Function Index (FFI), a questionnaire that informs us about the repercussion (pain, disability and restriction) that foot pathology has on the patient. It is made up of 23 items. The result is calculated using the following formula: sum of the questions / 230x100 = __%.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V Espí-López, Principal Investigator — University of Valencia
Locations (2):
- Spain (2):
  - Gemma V Espí López, Valencia
  - Gemma Victoria Espí-López, Valencia

IPD SHARING:
Plan to Share IPD: No